CLINICAL TRIAL: NCT05083299
Title: Multicenter, Therapeutic Use Observational Study to Evaluate the Effects of Concurrent Therapy of Sarpogrelate on Symptom Improvement in Patients With Peripheral Arterial Disease
Brief Title: Multicenter, Therapeutic Use Observational Study to Evaluate the Effects of Concurrent Therapy of Sarpogrelate
Status: Completed | Type: Observational
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Other Study IDs: DWAP_P401
Record Dates: First submitted 2021-10-06; First posted 2021-10-19 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Chronic Occlusive Arterial Disease
MeSH Terms: interventions — sarpogrelate

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Anpl-one SR Tablet: Patients who prescribed Anpl-one SR Tablet
  Interventions: Drug: Sarpogrelate

INTERVENTIONS:
Drug: Sarpogrelate — Anpl-one SR
  Other Names: Anpl-one SR

SUMMARY:
The study will evaluate the effect of Anpl-one SR Tablet on the improvement of symptoms in daily care environments using PAQ.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effect of Anple-one SR Tablet on the improvement of symptoms in daily care environments within the scope of 300 milligrams of Anpl-one SR Tablet (sarpogrelate hydrochloride agent) using PAQ.

ELIGIBILITY:
Inclusion Criteria:

1. Adults over 19 and under 80 years of age.
2. Patients who first administered Sarpogrelate hydrochloride drugs or less than 3 months to improve ischemic symptoms such as ulcers, pain, and coldness caused by chronic arterial obstruction (Burger's disease, obstructive arteriosclerosis, diabetic peripheral angiopathy, etc.).
3. Patient who voluntarily signed a written consent form approved by the Clinical Trial Review Committee or Ethics Committee and agreed to participate in the study by the patient or the subject's agent.

Exclusion Criteria:

1. Patient who is expected to have less than two years of life expectancy.
2. Patient who have bleeding within a week of participation in the study
3. Patient suffering from diseases that may increase bleeding during study participation (hemophilia, capillary placebo, digestive tube ulcer, urinary tract bleeding, hemoptysis, hyperself-bleeding, etc.).
4. A female patient who is likely to be pregnant or pregnant.
5. Female patients who are lactating or are scheduled to be lactated at the time of participation in the study.
6. Patients with severe renal disease and liver disease.

Ages: 19 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: As a result of the calculation for the number of survey subjects in this study, a total of 1507 subjects are required, and a total of 1,884 subjects are planned to be recruited in consideration of the dropout rate of 20%.
Sampling Method: Probability Sample
Enrollment: 1003 (Actual)
Dates: Start 2020-01-28 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
Change in Peripheral Artery Questionnaire | 24 weeks
  Change in Peripheral Artery Questionnaire at 24 weeks compared to baseline

SECONDARY OUTCOMES:
Peripheral Artery Questionnaire change | 12 weeks
  Peripheral Artery Questionnaire change at 12 weeks compared to baseline
Peripheral Artery Questionnaire change | 24 weeks
  Peripheral Artery Questionnaire change at 24 weeks compared to baseline
Change in each domain of Peripheral Artery Questionnaire | 24 weeks
  Change in each domain of Peripheral Artery Questionnaire at 24 weeks compared to baseline
Confirm the relationship between the ABI criteria and PAQ related to the diagnosis of PAD patients | 12 weeks
  Confirm the relationship between the ABI criteria and PAQ related to the diagnosis of PAD patients at 12 weeks
Confirm the relationship between the ABI criteria and PAQ related to the diagnosis of PAD patients | 24 weeks
  Confirm the relationship between the ABI criteria and PAQ related to the diagnosis of PAD patients at 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: BuKyung Kim, Principal Investigator — Kosin University Hospital
Locations (1):
- BuKyung Kim, Busan, South Korea

IPD SHARING:
Plan to Share IPD: No